CLINICAL TRIAL: NCT00017771
Title: A Pathophysiologic Study of Development of Distal Symmetrical Polyneuropathy in Individuals With Advanced HIV-1 Infection and Prior Antiretroviral Exposure
Brief Title: Nerve Damage in Patients With HIV Infection Who Have Been Treated With Anti-HIV Drugs
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: A5117; AACTG A5117; ACTG A5117; 10935 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2001-06-11; First posted 2001-08-31 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections; Peripheral Nervous System Disease
Keywords: HIV-1; CD4 Lymphocyte Count; Risk Factors; Hydroxyurea; Disease Progression; Alcohol Drinking; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Polyneuropathies; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases; Disease Progression; Alcohol Drinking; Polyneuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection

SUMMARY:
The purpose of this study is to find out what might increase nerve damage in people with HIV who have taken drugs for treatment of HIV disease. Another purpose is to see if nerve exams are done correctly before clinical research sites enroll HIV-infected patients.

Nerve damage is common in patients with HIV infection and can cause serious problems. The factors that place patients at risk are not well understood. This study will examine these factors in patients with advanced HIV infection and who have been taking anti-HIV drugs.

DETAILED DESCRIPTION:
Neurological complications in HIV infection are common and are significant sources of mortality and morbidity. The associated risk factors have not been clearly defined. Several studies have patients who are suited for analysis of peripheral neuropathy and can address the important clinical question of when a subject with asymptomatic neuropathy is most at risk for progressing to painful neuropathy. Some patients in this population with advanced HIV disease will likely have asymptomatic peripheral neuropathy at baseline, and will present an excellent opportunity for prospective study. Detailed quantitative assessments will be carried out to determine the incidence and course of peripheral neuropathy in this population. Risk factors for the development of new peripheral neuropathy, worsening of existing neuropathy, and progression to symptomatic peripheral neuropathy, such as CD4+ cell counts, HIV-1 viral load, and prior nucleoside analogue use, will be evaluated. The potential additive neurotoxic effects of hydroxyurea exposure in this population can also be analyzed.

HIV-infected patients are characterized for the presence or absence of neuropathy at [AS PER AMENDMENT 03/05/02: screening], baseline, Week 24, and Week 48. Entry variables are analyzed to determine predictors of progression from asymptomatic to symptomatic neuropathy or for worsening of symptomatic neuropathy. HIV-uninfected control volunteers have 1 visit [AS PER AMENDMENT 03/05/02: or 2 visits] for nerve conduction and Quantitative Sensory Testing (QST) evaluations to demonstrate proficiency with the testing methods prior to the enrollment of HIV-infected patients. HIV-infected patients are evaluated with the components of the Total Neuropathy Score (TNS) which includes signs (motor function, sensory function, and reflexes), symptoms (motor symptoms and sensory symptoms), QST (CASE IV - vibratory, cooling, and heat pain thresholds), and nerve conduction studies (sural nerve and peroneal nerve). Other evaluations include the Gracely Pain Scale and Visual Analog Scale pain diaries, paired skin biopsies from the right thigh and distal leg (total of 2), and peripheral blood lymphocyte analysis for quantitation of mitochondrial DNA content at entry and final study visit.

ELIGIBILITY:
Inclusion Criteria

Control volunteers will be eligible for this study if they:

* Are HIV negative.
* Are at least 18 years old.

Patients will be eligible for this study if they:

* Are HIV positive.
* Are at least 13 years old and can provide written consent from parent or guardian if under 18 years of age.
* Have taken anti-HIV drugs for at least 15 straight weeks any time in the past.
* Have a CD4 count of less than 300 cells/mm3.

Exclusion Criteria

Control volunteers will not be eligible for this study if they:

* Have any nerve-related problems.
* Have diabetes and nerve damage related to diabetes.
* Have long-term illness the doctor feels would interfere with the study.

Patients will not be eligible for this study if they:

* Have had spinal surgery.
* Have taken insulin or oral hypoglycemic products for diabetes mellitus within 30 days prior to study entry. Dietary control for diabetes is allowed.
* Have nerve damage related to diabetes.
* Have a nerve condition unrelated to HIV infection or antiretroviral therapy.
* Have alcohol-related medical complications within 6 months of study entry.
* Have vitamin B12 levels of less than 200 pg/ml or a history of vitamin B12 deficiency.

This study has been changed to modify the exclusion criteria. Earlier versions did not include some of these exclusion criteria.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected individuals who have previously undergone HIV treatment. HIV-uninfected to be used as controls.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2001-06; Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Simpson, Study Chair
Locations (18):
- United States (18):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Hawaii, Honolulu, Hawaii
  - The CORE Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Washington Univ / St Louis Connect Care, St Louis, Missouri
  - Washington Univ School of Medicine, St Louis, Missouri
  - Beth Israel Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Mount Sinai Med Ctr, Pittsburgh, Pennsylvania
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Result] Simpson DM, Kitch D, Evans SR, McArthur JC, Asmuth DM, Cohen B, Goodkin K, Gerschenson M, So Y, Marra CM, Diaz-Arrastia R, Shriver S, Millar L, Clifford DB; ACTG A5117 Study Group. HIV neuropathy natural history cohort study: assessment measures and risk factors. Neurology. 2006 Jun 13;66(11):1679-87. doi: 10.1212/01.wnl.0000218303.48113.5d. PMID 16769940
- [Derived] Roda RH, Bargiela D, Chen W, Perry K, Ellis RJ, Clifford DB, Bharti A, Kallianpur AR, Oliveira MF, Diaz MM, Rubin LH, Gavegnano C, McArthur JC, Hoke A, Polydefkis M. Large Mitochondrial DNA Deletions in HIV Sensory Neuropathy. Neurology. 2021 Jul 13;97(2):e156-e165. doi: 10.1212/WNL.0000000000012142. Epub 2021 May 4. PMID 33947785